CLINICAL TRIAL: NCT00059839
Title: A Phase III Trial of Treatment of Advanced-Stage Anaplastic Large Cell Lymphoma (ALCL) With Standard APO (Doxorubicin, Prednisone, Vincristine) Versus Consolidation With a Regimen Including Vinblastine
Brief Title: Comparison of Two Combination Chemotherapy Regimens With Either Vincristine or Vinblastine in Treating Patients With Advanced Anaplastic Large Cell Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANHL0131; CDR0000298777 (Other: Clinical Trials.gov); COG-ANHL0131 (Other: Children's Oncology Group)
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Results first posted 2013-10-08 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Lymphoma
Keywords: anaplastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large-Cell, Anaplastic | interventions — Doxorubicin; Mercaptopurine; Methotrexate; Prednisone; Vinblastine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard APO with Vincristine (Arm I ) (Experimental): In courses 1-3, patients receive doxorubicin hydrochloride (30 mg/m2) IV over 15 minutes, vincristine sulfate (1.5 mg/m2 (maximum dose 2 mg)) IV, and methotrexate intrathecally (age-adjusted dosing) (IT) on day 1 and oral prednisone (40 mg/m2/day) three times daily and oral mercaptopurine (225 mg/m2) once daily on days 1-5. In courses 4 and 5, patients receive doxorubicin (30 mg/m2), vincristine sulfate (1.5 mg/m2 (Maximum dose 2 mg)), prednisone (120 mg/m2/day), and mercaptopurine (225 mg/m2) as in courses 1-3. In courses 6-15, patients receive vincristine sulfate (1.5 mg/m2), prednisone (120 mg/m2/day), and mercaptopurine (225 mg/m2) as in courses 1-3 and methotrexate (60 mg/m2) IV on day 1. Treatment repeats every 21 days for up to 15 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: doxorubicin hydrochloride; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: vincristine sulfate
- Consolidation with Vinblastine (Experimental): In courses 1-3, patients receive doxorubicin hydrochloride (30 mg/m2) IV, methotrexate (age adjusted dosing) IT, prednisone (120 mg/m2/day), and mercaptopurine (225 mg/m2) as in arm I and vinblastine sulfate (4 mg/m2) IV over 1 minute on days 1, 8, and 15. In courses 4 and 5, patients receive doxorubicin hydrochloride (30 mg/m2) IV, prednisone (120 mg/m2/day), and mercaptopurine (225 mg/m2) as in arm I and vinblastine sulfate (4 mg/m2) as in arm II (courses 1-3). In courses 6-15, patients receive prednisone (120 mg/m2/day) and mercaptopurine (225 mg/m2) as in arm I, vinblastine sulfate (4 mg/m2) IV as in arm II (courses 1-3), and methotrexate (60 mg/m2) IV on day 1. Treatment repeats every 21 days for up to 15 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: doxorubicin hydrochloride; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: vinblastine sulfate

INTERVENTIONS:
Drug: doxorubicin hydrochloride — Given IV
Drug: mercaptopurine — Given by mouth
Drug: methotrexate — Given IV and intrathecally
Drug: prednisone — Given by mouth
Drug: vinblastine sulfate — Given IV
  Arms: Consolidation with Vinblastine
Drug: vincristine sulfate — Given IV
  Arms: Standard APO with Vincristine (Arm I )

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells. It is not yet known if combination chemotherapy with vinblastine is more effective than combination chemotherapy with vincristine in treating advanced anaplastic large cell lymphoma.

PURPOSE: Randomized phase III trial to compare the effectiveness of two combination chemotherapy regimens with either vinblastine or vincristine in treating patients who have newly diagnosed advanced anaplastic large cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of a consolidation chemotherapy regimen comprising doxorubicin and prednisone in combination with vincristine vs vinblastine, in terms of event-free survival, in patients with advanced anaplastic large cell lymphoma.
* Compare overall survival of patients treated with these regimens.
* Compare the toxic effects of these regimens in these patients.
* Correlate biological tumor characteristics and outcome in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study.

Patients are randomized at enrollment to receive either Standard APO regimen or a consolidation regimen including vinblastine (VBL).

* Induction therapy: All Patients receive doxorubicin IV over 15 minutes on days 1 and 22; vincristine IV on days 1, 8, 15, 22, and 29; oral prednisone 3 times daily on days 1-28; and intrathecal (IT) methotrexate on days 1, 8, and 22 (patients with central nervous system (CNS) disease at diagnosis receive additional methotrexate IT on days 15, 29, and 36).

Patients undergo restaging after Induction such that consolidation therapy is started on day 43. All patients with complete response (CR), complete response unconfirmed (CRu) or partial response (PR) proceed to Consolidation based on CT or MRI scans at the end of induction (week 6). All other patients will be removed from protocol therapy and will be followed until they meet the criteria for off study. Follow-up data will be required unless consent is withdrawn.

* Standard APO (Arm I): Patients receive course-specific regimens without vinblastine.

  * Courses 1-3: Patients receive doxorubicin IV over 15 minutes, vincristine IV, and methotrexate IT on day 1 and oral prednisone three times daily and oral mercaptopurine once daily on days 1-5.
  * Courses 4-5: Patients receive doxorubicin, vincristine, prednisone, and mercaptopurine as in courses 1-3.
  * Courses 6-15: Patients receive vincristine, prednisone, and mercaptopurine as in courses 1-3 and methotrexate IV on day 1.
* Consolidation with vinblastine (Arm II): Patients receive course-specific regimens including vinblastine.

  * Courses 1-3: Patients receive doxorubicin, methotrexate IT, prednisone, and mercaptopurine as in arm I and vinblastine IV over 1 minute on days 1, 8, and 15.
  * Courses 4-5: Patients receive doxorubicin, prednisone, and mercaptopurine as in arm I and vinblastine as in arm II (courses 1-3).
  * Courses 6-15: Patients receive prednisone and mercaptopurine as in arm I, vinblastine as in arm II (courses 1-3), and methotrexate IV on day 1.

In both arms and all courses, treatment repeats every 21 days for up to 15 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed monthly for 1 year, every 3 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 200-250 patients (100-125 per treatment arm) will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed advanced anaplastic large cell lymphoma

  * Cluster of differentiation antigen 30 (CD30+)
  * Murphy stage III or IV
* No B-cell large cell lymphoma
* No disease limited to the skin (regardless of how wide-spread)

PATIENT CHARACTERISTICS:

Age

* Under 21

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST) or alanine transaminase (ALT) less than 2.5 times ULN (unless due to lymphoma)

Renal

* Not specified

Cardiovascular

* Shortening fraction (SF) at least 27% by echocardiogram OR
* Ejection fraction (EF) at least 50% by radionuclide angiogram

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Prior steroids for management of a mediastinal mass allowed

Radiotherapy

* Prior limited-dose radiotherapy for a mediastinal mass allowed

Surgery

* Not specified

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 129 (Actual)
Dates: Start 2003-11; Primary Completion 2009-12 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Kraveka, DO, Study Chair — Medical University of South Carolina
Locations (159):
- United States (136):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital of Orange County, Orange, California
  - Sutter Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center - Oakland, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - Children's Hospital Center for Cancer and Blood Disorders, Aurora, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Simmons Cooper Cancer Institute, Springfield, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Floating Hospital for Children at Tufts - New England Medical Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Baystate Regional Cancer Program at D'Amour Center for Cancer Care, Springfield, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Children's Mercy Hospital, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Children's Hospital, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Overlook Hospital, Morristown, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Brooklyn Hospital Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Toledo Hospital, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Oregon Health and Science University Cancer Institute, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - T.C. Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine - Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Carilion Medical Center for Children at Roanoke Community Hospital, Roanoke, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center - Tacoma, Tacoma, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Midwest Children's Cancer Center at Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Westmead Institute for Cancer Research at Westmead Hospital, Westmead, New South Wales
  - Royal Children's Hospital, Brisbane, Queensland
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (16):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
  - Centre Hospitalier Universitaire de Quebec, Québec
- San Jorge Children's Hospital, Santurce, Puerto Rico
- Switzerland (3):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Swiss Pediatric Oncology Group Geneva, Geneva
  - Swiss Pediatric Oncology Group Lausanne, Lausanne

REFERENCES:
- [Derived] Alexander S, Kraveka JM, Weitzman S, Lowe E, Smith L, Lynch JC, Chang M, Kinney MC, Perkins SL, Laver J, Gross TG, Weinstein H. Advanced stage anaplastic large cell lymphoma in children and adolescents: results of ANHL0131, a randomized phase III trial of APO versus a modified regimen with vinblastine: a report from the children's oncology group. Pediatr Blood Cancer. 2014 Dec;61(12):2236-42. doi: 10.1002/pbc.25187. Epub 2014 Aug 23. PMID 25156886

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a multi-center, phase III, randomized trial for newly diagnosed children with advanced-stage anaplastic large cell lymphoma (ALCL). The study was activated on November 3, 2003 and the first date of enrollment was January 13, 2004.
Pre-assignment Details: Randomization occurs at the time of enrollment with all participants receiving Standard Induction of Doxorubicin, Prednisone and Vincristine (APO) and are evaluated at week 6 for continuation therapy.
Groups:
- Standard (APO) With Vincristine (Arm I): In courses 1-3, patients receive doxorubicin hydrochloride (30 mg/m2) IV over 15 minutes, vincristine sulfate (1.5 mg/m2 (maximum dose 2 mg)) IV, and methotrexate intrathecally (age-adjusted dosing) (IT) on day 1 and oral prednisone (40 mg/m2/day) three times daily and oral mercaptopurine (225 mg/m2) once daily on days 1-5. In courses 4 and 5, patients receive doxorubicin (30 mg/m2), vincristine sulfate (1.5 mg/m2 (Maximum dose 2 mg)), prednisone (120 mg/m2/day), and mercaptopurine (225 mg/m2) as in courses 1-3. In courses 6-15, patients receive vincristine sulfate (1.5 mg/m2), prednisone (120 mg/m2/day), and mercaptopurine (225 mg/m2) as in courses 1-3 and methotrexate (60 mg/m2) IV on day 1. Treatment repeats every 21 days for up to 15 courses in the absence of disease progression or unacceptable toxicity.
- Consolidation (Includes Vinblastine) (Arm II): In courses 1-3, patients receive doxorubicin hydrochloride (30 mg/m2) IV, methotrexate (age adjusted dosing) IT, prednisone (120 mg/m2/day), and mercaptopurine (225 mg/m2) as in arm I and vinblastine sulfate (4 mg/m2) IV over 1 minute on days 1, 8, and 15. In courses 4 and 5, patients receive doxorubicin hydrochloride (30 mg/m2) IV, prednisone (120 mg/m2/day), and mercaptopurine (225 mg/m2) as in arm I and vinblastine sulfate (4 mg/m2) as in arm II (courses 1-3). In courses 6-15, patients receive prednisone (120 mg/m2/day) and mercaptopurine (225 mg/m2) as in arm I, vinblastine sulfate (4 mg/m2) IV as in arm II (courses 1-3), and methotrexate (60 mg/m2) IV on day 1. Treatment repeats every 21 days for up to 15 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Standard (APO) With Vincristine (Arm I) | Consolidation (Includes Vinblastine) (Arm II)
Started | 65 | 64
Completed | 53 | 47
Not Completed | 12 | 17
Not completed — Death | 1 | 1
Not completed — Lack of Efficacy | 6 | 5
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 1 | 2
Not completed — Withdrawal by Subject | 1 | 6
Not completed — Ineligible | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard (APO) With Vincristine (Arm I) | Consolidation (Includes Vinblastine) (Arm II) | Total
Number analyzed (Participants) | 65 | 64 | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 62 | 62 | 124
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 27 | 51
  Male | 41 | 37 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 8 | 18
  Not Hispanic or Latino | 52 | 55 | 107
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 12 | 19
  White | 47 | 42 | 89
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 59 | 52 | 111
  Canada | 3 | 9 | 12
  Australia | 2 | 2 | 4
  Switzerland | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS)
Description: Percentage of EFS patients. This is measured as the time from study entry until disease progression, disease recurrence, occurrence of a second malignant neoplasm, or death from any cause. To measure Event Free Survival, repeated one-sided logrank tests will be performed The upper critical values are based on the one-sided alpha-spending functions of t2 (alpha=0.05) and the lower critical values are based on testing the alternative hypothesis at 0.005 level.
Time Frame: From first enrollment up to 3 years.
Population: 64 patients from Arm I were analyzed for this outcome measure, one patient was deemed ineligible. 61 patients from Arm II were analyzed for this outcome measure, three patients were deemed ineligible.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Standard (APO) With Vincristine (Arm I) | Consolidation (Includes Vinblastine) (Arm II)
Number analyzed (Participants) | 64 | 61
percentage of participants | 74 [61 to 84] | 79 [65 to 87]

ADVERSE EVENTS:
Description: 64 patients are included for Arm I adverse events as one patient was deemed ineligible. 61 patients are included for Arm II adverse events as three patients were deemed ineligible.
Arm/Group | Standard (APO) With Vincristine (Arm I) | Consolidation (Includes Vinblastine) (Arm II)
Serious Adverse Events (participants affected / at risk) | 2/64 | 4/61
Other Adverse Events (participants affected / at risk) | 47/64 | 52/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Standard (APO) With Vincristine (Arm I) (N=64) | Consolidation (Includes Vinblastine) (Arm II) (N=61)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
"Blood and lymphatic system disorders - Other" (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
"Cardiac disorders - Other" (Cardiac disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death NOS (General disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1/1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
CPK increased (Investigations) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
"Nervous system disorders - Other" (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard (APO) With Vincristine (Arm I) (N=64) | Consolidation (Includes Vinblastine) (Arm II) (N=61)
Anemia (Blood and lymphatic system disorders) | 14 (14) | 24 (24)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (7) | 18 (18)
"Cardiac disorders - Other" (Cardiac disorders) | 2 (2) | 0 (0)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 3 (3)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
"Eye disorders - Other" (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 5 (5)
Anal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 5 (5)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
"Gastrointestinal disorders - Other" (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 6 (6) | 7 (7)
Nausea (Gastrointestinal disorders) | 3 (3) | 8 (8)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 10 (10)
Chills (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 3 (3)
Fatigue (General disorders) | 3 (3) | 5 (5)
Fever (General disorders) | 4 (4) | 6 (6)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Irritability (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 3 (3) | 6 (6)
Catheter related infection (Infections and infestations) | 4 (4) | 1 (1)
Gum infection (Infections and infestations) | 0 (0) | 1 (1)
"Infections and infestations - Other" (Infections and infestations) | 6 (6) | 20 (20)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Penile infection (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
"Injury, poisoning and procedural complications - Other" (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 15 (15) | 26 (26)
Aspartate aminotransferase increased (Investigations) | 7 (7) | 16 (16)
Blood bilirubin increased (Investigations) | 2 (2) | 4 (4)
Creatinine increased (Investigations) | 1 (1) | 3 (3)
GGT increased (Investigations) | 3 (3) | 2 (2)
INR increased (Investigations) | 0 (0) | 1 (1)
"Investigations - Other" (Investigations) | 2 (2) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2) | 8 (8)
Neutrophil count decreased (Investigations) | 34 (34) | 47 (47)
Platelet count decreased (Investigations) | 6 (6) | 9 (9)
Serum amylase increased (Investigations) | 1 (1) | 1 (1)
Weight gain (Investigations) | 2 (2) | 2 (2)
Weight loss (Investigations) | 0 (0) | 3 (3)
White blood cell decreased (Investigations) | 20 (20) | 31 (31)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (8) | 9 (9)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3) | 6 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (5) | 12 (12)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 7 (7) | 12 (12)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4) | 6 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (4) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
"Musculoskeletal and connective tissue disorder - Other, specify" (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 9 (9)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 6 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3) | 7 (7)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Personality change (Psychiatric disorders) | 1 (1) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
"Respiratory, thoracic and mediastinal disorders - Other" (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
"Skin and subcutaneous tissue disorders - Other" (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 6 (6)
Hypotension (Vascular disorders) | 1 (1) | 4 (4)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No